CLINICAL TRIAL: NCT04191174
Title: Prevalence and Clinical Relevance of Ventilation Heterogeneity and Luminal Cellular Inflammation in Lung Cancer Patients Prior to Lung Resection
Brief Title: Ventilation Heterogeneity Prior to Lung Resection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: McMaster University (Other)
Collaborators: Cyclomedica Australia Pty Ltd (Unknown); Ontario Lung Association (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Other Study IDs: FIRH_Xe004
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: lung cancer; lung resection; ventilation heterogeneity; Technegas V SPECT; hyperpolarized 129Xe MRI; airway inflammation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults undergoing lung resection for lung cancer
  Interventions: Other: Hyperpolarized 129Xe MRI; Other: Technegas V SPECT; Other: Sputum Induction

INTERVENTIONS:
Other: Hyperpolarized 129Xe MRI — Hyperpolarized 129Xe MRI to evaluate ventilation heterogeneity
Other: Technegas V SPECT — Technegas V SPECT to evaluate ventilation heterogeneity
Other: Sputum Induction — Sputum induction to evaluate luminal cellular inflammation

SUMMARY:
This is a single centre prospective six-week observational study to understand the prevalence and clinical relevance of abnormal ventilation of the lung (assessed by Technegas ventilation single photon emission computed tomography (V SPECT) and hyperpolarized 129Xe magnetic resonance imaging (MRI)), in the presence or absence of airway inflammation (assessed by sputum cell counts), in lung cancer patients prior to lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing lung resection for lung cancer at St. Joseph's Healthcare (Hamilton, Ontario) in accordance with British Thoracic Society guidelines.
* Males and females ≥ 18 years of age.
* Able and willing to provide written informed consent.
* Able and willing to comply with the study protocol.

Exclusion Criteria:

* Previous lung resection surgery.
* Previous chest radiation.
* Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples.
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing lung resection (at St. Joseph's Healthcare Hamilton) for lung cancer as part of their clinical care
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Abnormal ventilation heterogeneity assessed by Technegas V SPECT | Baseline
  Proportion of patients with abnormal ventilation heterogeneity, assessed by Technegas V SPECT, prior to lung resection for lung cancer.
Abnormal ventilation heterogeneity assessed by 129Xe MRI | Baseline
  Proportion of patients with abnormal ventilation heterogeneity, assessed by 129Xe MRI, prior to lung resection for lung cancer.

SECONDARY OUTCOMES:
Technegas V SPECT ventilation heterogeneity and luminal cellular inflammation | Baseline
  Proportion of patients with preoperative luminal cellular inflammation in the preoperative ventilation heterogeneity normal and abnormal groups, assessed by Technegas V SPECT.
129Xe MRI ventilation heterogeneity and luminal cellular inflammation | Baseline
  Proportion of patients with preoperative luminal cellular inflammation in the preoperative ventilation heterogeneity normal and abnormal groups, assessed by 129Xe MRI.
Incidence of post-operative pulmonary complications (PPC): Technegas V SPECT ventilation heterogeneity | up to 4 weeks
  Difference in incidence of PPC and related impact measures in preoperative ventilation heterogeneity normal and abnormal patients, assessed by Technegas V SPECT
Incidence of PPC: 129Xe MRI ventilation heterogeneity | up to 4 weeks
  Difference in incidence of PPC and related impact measures in preoperative ventilation heterogeneity normal and abnormal patients, assessed by 129Xe MRI.
Incidence of PPC: Technegas V SPECT ventilation heterogeneity and luminal cellular inflammation | up to 4 weeks
  Difference in incidence of PPC and related impact measures in preoperative ventilation heterogeneity abnormal patients, assessed by Technegas V SPECT, with and without preoperative luminal cellular inflammation.
Incidence of PPC: 129Xe MRI ventilation heterogeneity and luminal cellular inflammation | up to 4 weeks
  Difference in incidence of PPC and related impact measures in preoperative ventilation heterogeneity abnormal patients, assessed by 129Xe MRI, with and without preoperative luminal cellular inflammation.

OTHER OUTCOMES:
Correlation between ventilation heterogeneity quantified by Technegas V SPECT and 129Xe MRI | Baseline
  Univariate correlation between preoperative ventilation heterogeneity quantified by Technegas V SPECT and 129Xe MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute for Respiratory Health, Research - St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agostini P, Cieslik H, Rathinam S, Bishay E, Kalkat MS, Rajesh PB, Steyn RS, Singh S, Naidu B. Postoperative pulmonary complications following thoracic surgery: are there any modifiable risk factors? Thorax. 2010 Sep;65(9):815-8. doi: 10.1136/thx.2009.123083. PMID 20805178
- [Background] Lugg ST, Agostini PJ, Tikka T, Kerr A, Adams K, Bishay E, Kalkat MS, Steyn RS, Rajesh PB, Thickett DR, Naidu B. Long-term impact of developing a postoperative pulmonary complication after lung surgery. Thorax. 2016 Feb;71(2):171-6. doi: 10.1136/thoraxjnl-2015-207697. PMID 26769017
- [Background] Pike D, Kirby M, Guo F, McCormack DG, Parraga G. Ventilation heterogeneity in ex-smokers without airflow limitation. Acad Radiol. 2015 Aug;22(8):1068-78. doi: 10.1016/j.acra.2015.04.006. Epub 2015 May 23. PMID 26008133
- [Background] Sheikh K, Paulin GA, Svenningsen S, Kirby M, Paterson NA, McCormack DG, Parraga G. Pulmonary ventilation defects in older never-smokers. J Appl Physiol (1985). 2014 Aug 1;117(3):297-306. doi: 10.1152/japplphysiol.00046.2014. Epub 2014 Jun 5. PMID 24903918
- [Background] Bajc M, Chen Y, Wang J, Li XY, Shen WM, Wang CZ, Huang H, Lindqvist A, He XY. Identifying the heterogeneity of COPD by V/P SPECT: a new tool for improving the diagnosis of parenchymal defects and grading the severity of small airways disease. Int J Chron Obstruct Pulmon Dis. 2017 May 26;12:1579-1587. doi: 10.2147/COPD.S131847. eCollection 2017. PMID 28603413